CLINICAL TRIAL: NCT03369145
Title: Influence of High-fat Overfeeding on Circulating Hepatokine Concentrations: a Randomised Crossover Study
Brief Title: High-fat Overfeeding, Hepatokines and Appetite Regulation
Acronym: OVEREAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Nottingham Trent University (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Scott Willis, Principal Investigator, Loughborough University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: R17-P144
Record Dates: First submitted 2017-11-20; First posted 2017-12-11 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Insulin Resistance; Type2 Diabetes Mellitus; Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: Hepatokines; High Fat Diet; Glycaemic Control; Fibroblast Growth Factor 21; Leukocyte Cell-derived Chemotaxin 2; Fetuin-A; Appetite; Ghrelin; Peptide YY
MeSH Terms: conditions — Insulin Resistance; Non-alcoholic Fatty Liver Disease; Obesity | interventions — Diet, High-Fat

STUDY DESIGN:
Intervention Model Description: The study design is a randomised, controlled, crossover design in which participants undertake two 7-day dietary conditions in a randomised order with a three week washout period in between.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat diet (Experimental): Participants will consume a hypercaloric, high-fat diet. Participants will be provided with all the food during the week and will be instructed to consume all of the foods provided and no extra calorie containing food or drink. In the event of leftover food, participants will be asked to return the food for measurement and subsequent subtraction from their total energy intake.
  Interventions: Dietary Supplement: High-fat diet
- Control diet (No Intervention): Participants will consume their normal 'habitual' diet for seven days which will be compared to their habitual diet recorded by a three day food diary before commencing the two diets. Participants will be instructed to carry on as normal and eat their usual diet and this period will be used as a comparator to the high-fat diet. They will also be told to record their food intake for 3 days during the diet to quantify their control diet.

INTERVENTIONS:
Dietary Supplement: High-fat diet — The high-fat diet will provide 7 days of overfeeding comprising of: +50% extra calories above the daily required intake, 65% of which is fat.
  Arms: High-fat diet

SUMMARY:
The present study will investigate the effect of high-fat overfeeding on a group of liver-secreted proteins linked to worsened blood sugar control, as well as proteins involved in appetite control. Participants will consume both a high-fat diet, consisting of 50% extra calories above their daily required intake, and a control diet, consisting of their normal 'habitual' diet, with each diet lasting seven days. The diets will be undertaken in a randomised order, with a period of three weeks separating the two diets. Blood samples will be taken before and after each diet to measure blood sugar control. Further blood samples will also be taken 24 hours and 72 hours into each diet to see how levels of the liver and appetite-regulating proteins change over the course of the seven days.

It is expected that blood sugar control will be worsened by the high-fat diet and this will be accompanied by increases in levels of the liver-secreted proteins and an impaired release of the appetite-regulating proteins into the blood.

DETAILED DESCRIPTION:
In recent years, researchers have identified a number of liver-secreted proteins, termed "hepatokines", which are thought to play an important role in inter-organ crosstalk between the liver and other metabolically active tissues such as skeletal muscle and adipose tissue. Specifically, previous studies have demonstrated that hepatokines contribute to whole body glucose and lipid homeostasis through acting in an endocrine-like fashion. Understanding how circulating concentrations of these hepatokines can be manipulated in humans is essential, as impaired blood glucose and lipid control is a key feature of metabolic diseases, such as type 2 diabetes and non-alcoholic fatty liver disease.

Previous research at Loughborough University has found that acute high-fat overfeeding for up to seven days can impair glycaemic control; however, the exact mechanisms responsible for these detrimental changes are not fully understood. Based upon previous evidence that hepatokine production is nutritionally modulated, the investigators believe that changes in hepatokine production may play a role in the detrimental metabolic effects seen following short-term, high-fat overfeeding which has implications for long-term metabolic health.

Appetite regulation is also thought to play a role in the pathophysiology of obesity and insulin resistance, as the impaired secretion of several appetite regulatory hormones in both fasting and postprandial conditions has been observed in obesity, which is characterised by an chronic excessive energy intake. Therefore, the investigators are also interested to examine the appetite regulatory hormone response to short-term, high-fat overfeeding.

The present study is a randomised, controlled, crossover study in which twelve recreationally active, healthy males will consume both a hypercaloric, high-fat diet (consisting of 50% extra energy above the daily requirement, 65% of which is fat) and a control diet (the participants' habitual diet) in a randomised fashion. A three-week washout period will separate the two diets in order to remove any lasting effects confounding the subsequent diet.

Following a prescreening session in which anthropometric data will be collected, participants will commence their first dietary condition. An oral glucose tolerance test will be performed before and after the two diets to measure changes in glycaemic control/whole body insulin sensitivity. Further blood samples will be taken 24 hours and 72 hours after commencing the diets in order to observe the time course of any changes in circulating hepatokine and appetite hormone concentrations. Physical activity will also be monitored for the duration of the two dietary conditions to ensure that habitual physical activity levels are maintained.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active - ≤ 2 structured exercise sessions per week
* BMI between 18.5 - 27.9 kg/m2
* Body fat percentage < 20%
* Metabolically healthy - No known cardiovascular or metabolic disease such as diabetes, respiratory or heart disease.
* Non-smoker
* Weight stable in the past 6 months
* Normal fasting blood glucose levels (3.6 - 5.5 mmol/l)

Exclusion Criteria:

* Contraindications to exercise
* Needle Phobia

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Leukocyte cell-derived chemotaxin 2 (LECT2) | Baseline, 1 day, 3 days, 7 days
  Time-course of LECT2 plasma concentrations across the 7-day dietary interventions

SECONDARY OUTCOMES:
Fibroblast growth factor 21 (FGF21) | Baseline, 1 day, 3 days, 7 days
  Time-course of FGF21 plasma concentrations across the 7-day dietary interventions
Fetuin-A | Baseline, 1 day, 3 days, 7 days
  Time-course of Fetuin-A plasma concentrations across the 7-day dietary interventions
Acylated ghrelin | Baseline, 1 day, 3 days, 7 days
  Time-course of acylated ghrelin plasma concentrations across the 7-day dietary interventions
Peptide YY (PYY) | Baseline, 1 day, 3 days, 7 days
  Time-course of PYY plasma concentrations across the 7-day dietary interventions
C-Terminal Telopeptide of Type 1 Collagen (CTX) | Baseline, 1 day, 3 days, 7 days
  Time-course of CTX plasma concentrations across the 7-day dietary interventions
N-Terminal Propeptide of Type 1 Procollagen (P1NP) | Baseline, 1 day, 3 days, 7 days
  Time-course of P1NP plasma concentrations across the 7-day dietary interventions
Visual Analogue Scale for Subjective Ratings of Appetite | Baseline, 1 day, 3 days, 7 days
  Time-course of subjective ratings of hunger across the 7-day dietary interventions, measured using an appetite visual analogue scale. The scale is divided into subscales of different appetite perceptions including: hunger, fullness, satisfaction and prospective food consumption. Each subscale is rated on a 100mm scale (i.e. from 0 - 100), with a rating of 100 fully supporting the perception and a rating of 0 fully opposing the perception.
Subjective food preference | Baseline, 1 day, 3 days, 7 days
  Time-course of subjective food preference across the 7-day dietary interventions, measured using the Leeds Food Preference Questionnaire.
Whole-body insulin sensitivity | Baseline, 7 Days
  Changes in whole-body insulin sensitivity using the Matsuda Index, calculated from plasma glucose and insulin concentrations during the oral glucose tolerance test
Homeostasis model assessment of insulin resistance (HOMA-IR) | Baseline, 1 day, 3 days, 7 days
  Changes in HOMA-IR (a marker of hepatic insulin resistance) using baseline concentrations of plasma glucose and insulin.
Adipose tissue insulin resistance (ADIPO-IR) | Baseline, 1 day, 3 days, 7 days
  Changes in ADIPO-IR using baseline concentrations of plasma insulin and non-esterified free fatty acids.
Physical activity and sedentary behaviour | 7 days (per diet)
  Amounts of sitting time, standing time, light activity and moderate-vigorous activity will be measured across the duration of each diets to compare between the two. This will be Measured using Acitgraph and ActivPAL monitors.
Resting Metabolic Rate | Baseline, 7 Days
  Changes in resting metabolic rate in response to the diets will be measured using indirect calorimetry and estimated using the Haldane transformation.
Fat Oxidation | Baseline, 7 Days
  Changes in fat oxidation in response to the diets will be measured using indirect calorimetry and estimated using the Haldane transformation.
Blood pressure | Baseline, 1 day, 3 days, 7 days
  Changes in blood pressure (systolic and diastolic) across the two dietary interventions will be measured using an automated pressure cuff.
Body weight | Baseline, 1 day, 3 days, 7 days
  Changes in body weight across the two dietary interventions.
Body fat percentage | Baseline, 7 Days
  Changes in body fat percentage across the two dietary interventions using bioelectrical impedance analysis.

CONTACTS AND LOCATIONS:
Overall Officials: James A King, PhD, Principal Investigator — Loughborough University; Scott A Willis, MSc, Principal Investigator — Loughborough University
Locations (2):
- United Kingdom (2):
  - National Centre for Sport and Exercise Medicine, Loughborough University, Loughborough, Leicestershire
  - Clifton Campus, Nottingham Trent University, Nottingham, Nottinghamshire

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Badman MK, Pissios P, Kennedy AR, Koukos G, Flier JS, Maratos-Flier E. Hepatic fibroblast growth factor 21 is regulated by PPARalpha and is a key mediator of hepatic lipid metabolism in ketotic states. Cell Metab. 2007 Jun;5(6):426-37. doi: 10.1016/j.cmet.2007.05.002. PMID 17550778
- [Background] Dasgupta S, Bhattacharya S, Biswas A, Majumdar SS, Mukhopadhyay S, Ray S, Bhattacharya S. NF-kappaB mediates lipid-induced fetuin-A expression in hepatocytes that impairs adipocyte function effecting insulin resistance. Biochem J. 2010 Aug 1;429(3):451-62. doi: 10.1042/BJ20100330. PMID 20482516
- [Background] Groop LC. Insulin resistance: the fundamental trigger of type 2 diabetes. Diabetes Obes Metab. 1999 May;1 Suppl 1:S1-7. doi: 10.1046/j.1463-1326.1999.0010s1001.x. PMID 11220283
- [Background] Hulston CJ, Churnside AA, Venables MC. Probiotic supplementation prevents high-fat, overfeeding-induced insulin resistance in human subjects. Br J Nutr. 2015 Feb 28;113(4):596-602. doi: 10.1017/S0007114514004097. Epub 2015 Jan 29. PMID 25630516
- [Background] Lan F, Misu H, Chikamoto K, Takayama H, Kikuchi A, Mohri K, Takata N, Hayashi H, Matsuzawa-Nagata N, Takeshita Y, Noda H, Matsumoto Y, Ota T, Nagano T, Nakagen M, Miyamoto K, Takatsuki K, Seo T, Iwayama K, Tokuyama K, Matsugo S, Tang H, Saito Y, Yamagoe S, Kaneko S, Takamura T. LECT2 functions as a hepatokine that links obesity to skeletal muscle insulin resistance. Diabetes. 2014 May;63(5):1649-64. doi: 10.2337/db13-0728. Epub 2014 Jan 29. PMID 24478397
- [Background] Meex RCR, Watt MJ. Hepatokines: linking nonalcoholic fatty liver disease and insulin resistance. Nat Rev Endocrinol. 2017 Sep;13(9):509-520. doi: 10.1038/nrendo.2017.56. Epub 2017 Jun 9. PMID 28621339
- [Background] Parry SA, Smith JR, Corbett TR, Woods RM, Hulston CJ. Short-term, high-fat overfeeding impairs glycaemic control but does not alter gut hormone responses to a mixed meal tolerance test in healthy, normal-weight individuals. Br J Nutr. 2017 Jan;117(1):48-55. doi: 10.1017/S0007114516004475. Epub 2017 Jan 24. PMID 28115026
- [Background] Uebanso T, Taketani Y, Yamamoto H, Amo K, Ominami H, Arai H, Takei Y, Masuda M, Tanimura A, Harada N, Yamanaka-Okumura H, Takeda E. Paradoxical regulation of human FGF21 by both fasting and feeding signals: is FGF21 a nutritional adaptation factor? PLoS One. 2011;6(8):e22976. doi: 10.1371/journal.pone.0022976. Epub 2011 Aug 1. PMID 21829679
- [Background] Lean ME, Malkova D. Altered gut and adipose tissue hormones in overweight and obese individuals: cause or consequence? Int J Obes (Lond). 2016 Apr;40(4):622-32. doi: 10.1038/ijo.2015.220. Epub 2015 Oct 26. PMID 26499438
- [Derived] Willis SA, Sargeant JA, Yates T, Takamura T, Takayama H, Gupta V, Brittain E, Crawford J, Parry SA, Thackray AE, Varela-Mato V, Stensel DJ, Woods RM, Hulston CJ, Aithal GP, King JA. Acute Hyperenergetic, High-Fat Feeding Increases Circulating FGF21, LECT2, and Fetuin-A in Healthy Men. J Nutr. 2020 May 1;150(5):1076-1085. doi: 10.1093/jn/nxz333. PMID 31919514

DOCUMENTS (3):
  • Study Protocol (2017-11-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03369145/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03369145/SAP_001.pdf
  • Informed Consent Form (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03369145/ICF_002.pdf